CLINICAL TRIAL: NCT07185399
Title: Systems Biological Analysis of Immune Responses to RSV Vaccine
Acronym: RSV SB
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Open Philanthropy (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00010088
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: RSV vaccine; Lower respiratory track disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moderna RSV vaccine (MRESVIA) (Experimental): Adults who are ≥60 years of age and are eligible to receive FDA-approved RSV vaccines under standard clinical recommendations receive a single dose of the Moderna RSV vaccine (MRESVIA).
  Interventions: Biological: Moderna RSV vaccine

INTERVENTIONS:
Biological: Moderna RSV vaccine — Participants will receive the MRESVIA vaccine (Moderna RSV vaccine) as part of the study. The vaccine will be administered by trained clinical personnel at the Hope Clinic. MRESVIA is FDA-approved and will be used in accordance with its licensed indication for adults aged 60 years and older. MRESVIA is an mRNA-based RSV vaccine containing 50 micrograms (mcg) of nucleoside-modified mRNA encoding the RSV prefusion F glycoprotein. It is supplied as a frozen injectable suspension in single-dose, pre-filled syringes. The vaccine is administered as a single 0.5 milliliter (mL) intramuscular injection.

SUMMARY:
The purpose of this study is to characterize the immune response to the FDA-approved mRNA-based RSV vaccine in adults ≥60 years of age, using a systems biology approach. The study aims to generate high-resolution immunologic and systems biology data following vaccination to identify early biomarkers of response and gain mechanistic insight into host immunity.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is a leading cause of lower respiratory tract disease (LRTD) in older adults and individuals with chronic comorbidities. In response to this burden, several RSV vaccines have recently been licensed for use in adults ≥60 years of age, including products developed by Pfizer, GlaxoSmithKline (GSK), and Moderna. These vaccines represent distinct technological platforms - recombinant protein with adjuvant, bivalent prefusion F (preF) subunit, and messenger RNA (mRNA), respectively - each with demonstrated efficacy in large-scale clinical trials.

Understanding the immunological mechanisms and durability of protection across these platforms remains a major research priority, particularly given the increased use of next-generation vaccine technologies such as mRNA. Systems biology approaches, including transcriptomics, proteomics, metabolomics and advanced immune profiling, provide a powerful means to identify early biomarkers of immunogenicity and long-term antibody persistence. Such approaches have successfully revealed predictive immune signatures in response to a variety of vaccines.

In parallel studies, the researchers have collected samples from individuals who received the Pfizer and GSK RSV vaccines at retail pharmacies under routine clinical use. However, the mRNA-based RSV vaccine (MRESVIA, developed by Moderna) has been less widely deployed to date in community settings, limiting opportunities to collect samples prospectively under real-world conditions. As a result, the researchers are establishing this dedicated protocol to characterize the immune response to MRESVIA using a systems biology approach. Through comprehensive sampling at early and late timepoints post-vaccination, the researchers aim to define molecular and cellular features unique to the mRNA platform and identify early predictors of immune response magnitude and durability. These data will also support future cross-platform comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥60 years of age at the time of enrollment.
* Able and willing to provide written informed consent.
* Eligible for receipt of an FDA-approved RSV vaccine (MRESVIA) per Advisory Committee on Immunization Practices (ACIP)/Centers for Disease Control and Prevention (CDC) guidelines.
* Available for all study visits and procedures, including follow-up through Day 180.
* Willing to allow access to prior RSV vaccination history (if applicable) for eligibility verification

Exclusion Criteria:

* History of severe allergic reaction (e.g., anaphylaxis) to any prior vaccines or any component of the MRESVIA vaccine, including polyethylene glycol (PEG), the amino lipid SM-102 (SM-102), or other listed excipients.
* Acute illness or fever (temperature ≥100.4°F) at the time of vaccination (participant may be rescheduled).
* Immunocompromising conditions, including:

  * Current cancer chemotherapy or immunosuppressive therapy.
  * History of hematologic malignancies or other immune-mediated diseases that would interfere with vaccine response.
  * Known or suspected HIV infection with cluster of differentiation 4 (CD4) count <200 or uncontrolled viremia.
* Clinically significant cardiac, pulmonary, renal, hepatic, or neurological disease that, in the opinion of the investigator, would preclude participation or confound interpretation of immune data.
* Uncontrolled autoimmune disorder.
* Current use of systemic corticosteroids equivalent to ≥20 mg prednisone daily for more than 14 consecutive days in the past month.
* History of Guillain-Barré Syndrome or other demyelinating neurological disorders.
* History of myocarditis, pericarditis, or myopericarditis within the last 2 months.
* Any bleeding disorder that poses a risk for venipuncture or vaccination complications.
* Participation in another clinical trial involving an investigational agent within 30 days of enrollment.
* Receipt or plan receipt of vaccines in the past an upcoming 28 days.
* Prior receipt of any RSV vaccine.
* Receipt of blood products or immune globulin within the prior 3 months.
* History of excessive alcohol consumption or drug use, or psychiatric/social/occupational conditions that may interfere with study compliance.
* Any other condition that, in the opinion of the investigator, may interfere with study conduct or participant safety.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Antibody Titers | Days 28 and 180 post-vaccination
  The magnitude of RSV-specific antibody responses following vaccination with an mRNA RSV vaccine (MRESVIA) is assessed as antibody titers at Days 28 and 180 post-vaccination.

SECONDARY OUTCOMES:
Frequency of Grade 2 or Higher Adverse Events | Day 28 post-vaccination
  The frequency of unsolicited adverse events (AEs) of Grade 2 or higher occurring within 28 days following vaccination will be examined.
Severity of Grade 2 or Higher Adverse Events | Day 28 post-vaccination
  The severity of unsolicited adverse events (AEs) of Grade 2 or higher occurring within 28 days following vaccination will be examined.
Occurrence of Serious Adverse Events | Up to Day 180 post-vaccination
  The occurrence of any serious adverse event (SAE) at any point during the 6-month follow-up period will be examined.
Occurrence of Adverse Events Meeting VAERS Reporting Criteria | Up to Day 180 post-vaccination
  The occurrence of any adverse event that meets VAERS reporting criteria during the 6-month follow-up will be examined. VAERS reporting criteria include: Anaphylaxis (within 7 days); Syncope (within 7 days); Shoulder Injury Related to Vaccine Administration (SIRVA); Acute complications or sequelae of anaphylaxis, syncope, or SIRVA; Events listed as contraindications in the vaccine's package insert; Any SAE, especially if unexpected or deemed related to the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared upon reasonable request, following completion of primary analyses. Data that will be available for sharing include de-identified demographic, safety, and immunogenicity data, as well as omics datasets (e.g., transcriptomics, proteomics, metabolomics) collected pre- and post-vaccination. Data dictionaries will also be provided.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available within 12 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Data will be available for sharing with qualified researchers from academic, nonprofit, or governmental institutions, for the purposes of analyses consistent with advancing scientific knowledge in vaccinology and immunology. Requests will be reviewed by the study PI. Approved investigators will sign a data use agreement (DUA) and data will be shared through secure transfer methods.